CLINICAL TRIAL: NCT00972179
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AMG 157 in Healthy Subjects
Brief Title: Safety Study of Tezepelumab (AMG 157) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20080390
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2022-05-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers
MeSH Terms: interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: The cohorts will enroll sequentially: enrollment to the subsequent cohort (ie, next higher dose) will proceed only after the previous dose is determined to be safe and well tolerated by a blinded review of available safety data conducted on day 43 of the previous cohort. Within each dose cohort, participants will be randomized 3:1 to receive tezepelumab or placebo.
Who Masked: Participant, Investigator

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab will be administered subcutaneously (SC) at doses from 35 mg once every 28 days (Q28D) (cohort 1) up to 210 mg once every 7 days (Q7D) (cohort 5) and an intravenous (IV) dose cohort of 700 mg Q28D (cohort 6).
  Interventions: Drug: Tezepelumab
- Placebo (Placebo Comparator): Two participants in each cohort (cohorts 1 to 6) will receive matching placebo administered subcutaneously (cohorts 1-5) or intravenously (cohort 6), matching the treatment regiment of tezepelumab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Administered by subcutaneous or intravenous injection.
  Arms: Placebo
Drug: Tezepelumab — Administered by subcutaneous or intravenous injection
  Other Names: AMG 157; Tezspire
  Arms: Tezepelumab

SUMMARY:
The primary objective is to evaluate the safety, tolerability, and immunogenicity of multiple-dose administration of tezepelumab in healthy adults.

DETAILED DESCRIPTION:
This study will follow a randomized, multiple-dose, double-blind, placebo-controlled, sequential dose-escalation study design. The study will consist of five subcutaneous (SC) cohorts and one intravenous (IV) cohort. Each dose cohort is planned to enroll 8 participants, randomized such that 6 participants will receive tezepelumab and 2 will receive placebo (3:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign an Institutional Review Board (IRB) approved informed consent form before any study-specific procedures;
* Healthy subject, aged between 18 and 45 years, inclusive;
* Female subject must be of non-reproductive potential (ie, postmenopausal by history - no menses for ≥ 1 year and by follicle-stimulating hormone (FSH) [using local reference ranges]; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy);
* Male subjects with female partner of childbearing potential who agrees to inform their female partner of their participation in this clinical study and use highly effective methods of birth control during the study. (Highly effective methods of birth control may include abstinence, vasectomy, or a condom with spermicide in combination with either hormonal birth control, intra-uterine device, or barrier methods used by the woman);
* Male subject who agrees to use birth control for five months after last dose of study medication, male subject who agrees not to donate sperm during the study and for five months after last dose of study medication;
* Healthy subject with a body mass index (BMI) between 18 and 32 kg/m^2, inclusive at screening;
* Subject must have normal or clinically acceptable physical examination and electrocardiogram (ECG) results prior to Day 1 based on the opinion of the investigator;
* Subject must have normal or clinically acceptable clinical laboratory tests at screening as determined by Amgen and the investigator;
* Subject must have adequate renal function (defined as creatinine clearance > 80 mL/min using the Cockcroft Gault equation).

Exclusion Criteria:

* Subject who has history or evidence of a clinically significant disorder, condition or disease (including but not limited to cardiopulmonary, oncologic, immunologic, autoimmune, collagen vascular, renal, metabolic, hematologic or psychiatric), that, in the opinion of the Investigator in consultation with the Amgen physician, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* Subject who has evidence of any active or suspected bacterial, viral, fungal or parasitic infections within the past 30 days prior to randomization (eg, common cold, viral syndrome, flu-like symptoms). Subject who, in the opinion of the investigator, has a high risk of parasitic disease is also excluded;
* Subject who has known positive tuberculin skin test (if not treated with appropriate chemoprophylaxis) or recent (within six months from randomization) exposure to an individual with active tuberculosis;
* Subject who has history of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers within five years before randomization of the study;
* Subject who has known type I/II diabetes;
* Subject who uses nonprescription drugs within 14 days prior to randomization and for the entire duration of the study. All herbal supplements, vitamins, and nutritional supplements taken within the last 30 days prior to dosing on Day 1 (and continued use, if appropriate), must be reviewed and approved by the PI and Amgen Medical Monitor;
* Subject who has used any systemic cytotoxic or systemic immunosuppressive medications (other than corticosteroids) within 6 months prior to randomization and for the entire duration of the study or has used any corticosteroid, topical cytotoxic or topical immunosuppressive medications within 30 days or five half-lives (whichever is longer) prior to randomization and for the entire duration of the study;
* Subject who has previously received any other therapeutic monoclonal antibody;
* Subject who has previously received any investigational drug (or is currently using an investigational device) within 30 days or five half-lives (whichever is longer) prior to randomization;
* Subject who has tested positive for drugs and/or alcohol use at screening or before randomization, subject who has consumed alcohol within 48 hours prior to any study visit including screening, and subject with alcohol intake of > 2 drinks/day on average during the study (one drink being equivalent to 12 ounces of regular beer, 8 to 9 ounces of malt liquor, 5 ounces of wine or 1.5 ounces of 80 proof distilled spirits);
* Female subject who is pregnant or lactating; female subject who is of child-bearing potential;
* Subject who has donated blood (including blood products) or experienced loss of blood ≥ 500 mL within two months of study screening;
* Subject who is positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, or hepatitis C antibodies;
* Subject who has regularly used nicotine or tobacco containing products (including but not limited to: snuff, chewing tobacco, cigars, cigarettes, pipes, or nicotine patches) during six months before randomization and during the study;
* Subject who has any other condition that might reduce the chance of obtaining data (eg, known poor compliance) required by the protocol or that might compromise the ability to give truly informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09-15 (Actual); Primary Completion 2011-01-09 (Actual); Study Completion 2011-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Parnes JR, Sullivan JT, Chen L, Dias C. Pharmacokinetics, Safety, and Tolerability of Tezepelumab (AMG 157) in Healthy and Atopic Dermatitis Adult Subjects. Clin Pharmacol Ther. 2019 Aug;106(2):441-449. doi: 10.1002/cpt.1401. Epub 2019 Mar 23. PMID 30779339
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: Participants were enrolled into 1 of 6 cohorts. In the first 5 cohorts escalating subcutaneous doses of tezepelumab were compared with placebo and in cohort 6 a regimen of intravenous tezepelumab was compared with placebo. Within each cohort, healthy participants were randomized at a 6:2 ratio to receive either tezepelumab or placebo.
Groups:
- Tezepelumab 35 mg Q28D: Participants received 35 mg tezepelumab by subcutaneous injection once every 28 days (Q28D) for 3 doses.
- Tezepelumab 105 mg Q28D: Participants received 105 mg tezepelumab by subcutaneous injection once every 28 days for 3 doses.
- Tezepelumab 210 mg Q28D: Participants received 210 mg tezepelumab by subcutaneous injection once every 28 days for 3 doses.
- Tezepelumab 210 mg Q14D: Participants received 210 mg tezepelumab by subcutaneous injection once every 14 days (Q14D) for 6 doses.
- Tezepelumab 210 mg Q7D: Participants received 210 mg tezepelumab by subcutaneous injection once every 7 days (Q7D) for 12 doses.
- Tezepelumab 700 mg Q28D IV: Participants received 700 mg tezepelumab by intravenous injection once every 28 days for 3 doses.
- Placebo: Participants received matching placebo administered subcutaneously (Cohorts 1-5) or intravenously (Cohort 6), matching the treatment regimen of tezepelumab.
Period: Overall Study
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV | Placebo
Started | 6 | 6 | 6 | 6 | 7 | 6 | 12
Completed | 5 | 3 | 5 | 5 | 5 | 3 | 8
Not Completed | 1 | 3 | 1 | 1 | 2 | 3 | 4
Not completed — Noncompliance | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 1 | 0 | 0 | 2
Not completed — Administrative Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug (Safety population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 12 | 49
Age, Continuous [Mean (Standard Deviation); unit: year] | 29.8 (9.3) | 34.8 (5.8) | 32.3 (5.3) | 31.5 (5.6) | 36.1 (7.7) | 27.7 (4.1) | 34.1 (5.2) | 32.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 4 | 1 | 0 | 2 | 7
  Male | 6 | 6 | 6 | 2 | 6 | 6 | 10 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 0 | 2 | 1 | 4 | 3 | 4 | 17
  Black or African American | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Hispanic or Latino | 3 | 6 | 4 | 5 | 3 | 1 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Adverse events (AEs) include any untoward medical occurrence in a trial participant administered a study drug and does not necessarily have a causal relationship with this treatment. AEs include worsening of a pre-existing medical condition and laboratory value changes requiring therapy or adjustment in prior therapy.
  AEs were assessed for severity according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3, where Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = severe AE, Grade 4 = life-threatening AE and Grade 5 = death due to AE.
  Relationship to study treatment was determined by the investigator.
  A serious adverse event (SAE) is defined as an AE that met 1 or more of below criteria:
  * was fatal;
  * was life threatening;
  * required in-patient hospitalization or prolongation of existing hospitalization;
  * resulted in persistent or significant disability/incapacity;
  * was a congenital anomaly/birth defect;
  * other significant medical hazard.
Time Frame: From first dose of study drug up to day 169
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Tezepelumab 35 mg Q28D: Participants received 35 mg tezepelumab by subcutaneous injection once every 28 days (Q28D) for three doses.
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 12
Participants
  Any adverse event | 4 | 4 | 2 | 6 | 5 | 3 | 10
  Serious adverse events | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AE Leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE Leading to discontinuation from study | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 adverse events | 1 | 0 | 0 | 1 | 1 | 1 | 2
  Grade 4 adverse events | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Fatal (grade 5) adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any treatment-related adverse event | 2 | 0 | 1 | 1 | 3 | 0 | 2

2. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Tezepelumab
Description: The pharmacokinetic (PK) parameter Tmax was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The concentration of tezepelumab in human serum was measured using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification of the assay was 10 ng/ml.
Time Frame: First dose: Day 1 predose, end of infusion (EOI; IV cohort only), 4 hours, 3, 7, 14 (Q14D & Q28D only) and 28 days (Q28D only) postdose. Last Dose: Day 57 (Q28D), Day 71 (Q14D) and Day 78 (Q7D) predose, EOI (IV cohort), 4 hours, 3, 7, 14, 28 days postdose
Population: Participants who received tezepelumab and had a sufficient number of serum concentration measurements for computing the PK parameter after first dose and after last dose.
Measure: Median (Full Range); unit: hours
Groups:
- Tezepelumab 105 mg Q28D: Participants received 105 mg tezepelumab by subcutaneous injection once every 28 days for three doses.
- Tezepelumab 210 mg Q28D: Participants received 210 mg tezepelumab by subcutaneous injection once every 28 days for three doses.
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6
hours
  First dose | 160 [69.7 to 167] | 71.5 [70.4 to 167] | 118 [68.7 to 166] | 70.7 [69.9 to 168] | 164 [66.9 to 165] | 4.00 [1.13 to 4.17]
  Last dose: number analyzed (Participants) | 5 | 3 | 5 | 6 | 5 | 5
  Last dose | 166 [68.6 to 176] | 71.8 [70.7 to 167] | 167 [69.3 to 168] | 66.5 [65.1 to 162] | 74.4 [65.9 to 164] | 3.97 [1.17 to 4.03]

3. Primary Outcome: Number of Participants Who Developed Anti-tezepelumab Antibodies After Initiation of Treatment
Description: All study samples (tezepelumab and placebo) were tested using an electrochemiluminescence (ECL) based immunoassay to detect and confirm the presence of antibodies capable of binding to tezepelumab. Samples identified as positive in the immunoassay were tested in a receptor-binding ECL-based assay to detect neutralizing or inhibitory effects toward tezepelumab.
  The number of participants with positive anti-tezepelumab binding antibodies / neutralizing antibodies at any time post-baseline with a negative or no result at baseline is reported.
Time Frame: For Q28D groups: Days 28, 56, 85, 113, and 169; For Q14D and Q7D groups: Days 29, 57, 85, 113, 141, and 169
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 12
Participants
  Anti-tezepelumab binding antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anti-tezepelumab neutralizing antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Tezepelumab
Description: The PK parameter Cmax was estimated based on the serum concentrations of tezepelumab using noncompartmental methods. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/ml.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6
µg/mL
  First dose | 3.70 (1.16) | 10.7 (3.13) | 23.6 (9.50) | 23.8 (5.40) | 18.0 (4.58) | 294 (48.2)
  Last dose: number analyzed (Participants) | 5 | 3 | 5 | 6 | 5 | 5
  Last dose | 6.29 (2.02) | 16.6 (2.02) | 37.4 (17.5) | 63.8 (13.5) | 117 (45.6) | 370 (74.9)

5. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUCtau) for Tezepelumab
Description: The PK parameter AUCtau was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The dosing interval (tau) was 28 days, 14 days or 7 days depending on the treatment arm.
  The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/ml.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7 | 6
days*µg/mL
  First dose | 78.9 (23.4) | 237 (50.5) | 481 (171) | 263 (49.2) | 84.3 (34.9) | 2980 (395)
  Last dose: number analyzed (Participants) | 5 | 3 | 5 | 6 | 5 | 5
  Last dose | 136 (35.9) | 333 (28.8) | 799 (338) | 787 (180) | 732 (224) | 4050 (1270)

6. Secondary Outcome: Accumulation Ratio Based on AUCtau
Description: Accumulation ratio (AR) based on AUCtau was calculated as AUCtau after last dose / AUCtau after first dose, except for the Q7D cohort where AR was calculated as AUCtau after last dose / area under the concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) after first dose.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV
Number analyzed (Participants) | 5 | 3 | 5 | 6 | 5 | 5
ratio | 1.82 (0.262) | 1.64 (0.0883) | 1.59 (0.242) | 2.89 (0.892) | 8.23 (1.93) | 1.34 (0.314)

7. Secondary Outcome: Accumulation Ratio Based on Cmax
Description: Accumulation ratio based on Cmax calculated as Cmax after last dose / Cmax after first dose
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV
Number analyzed (Participants) | 5 | 3 | 5 | 6 | 5 | 5
ratio | 1.79 (0.392) | 1.66 (0.0901) | 1.59 (0.288) | 2.84 (0.965) | 6.74 (1.69) | 1.30 (0.176)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to day 169
Groups:
- Tezepelumab Total: All participants who received tezepelumab.
Arm/Group | Tezepelumab 35 mg Q28D | Tezepelumab 105 mg Q28D | Tezepelumab 210 mg Q28D | Tezepelumab 210 mg Q14D | Tezepelumab 210 mg Q7D | Tezepelumab 700 mg Q28D IV | Tezepelumab Total | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 1/37 | 0/12
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/6 | 6/6 | 5/7 | 3/6 | 24/37 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tezepelumab 35 mg Q28D (N=6) | Tezepelumab 105 mg Q28D (N=6) | Tezepelumab 210 mg Q28D (N=6) | Tezepelumab 210 mg Q14D (N=6) | Tezepelumab 210 mg Q7D (N=7) | Tezepelumab 700 mg Q28D IV (N=6) | Tezepelumab Total (N=37) | Placebo (N=12)
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tezepelumab 35 mg Q28D (N=6) | Tezepelumab 105 mg Q28D (N=6) | Tezepelumab 210 mg Q28D (N=6) | Tezepelumab 210 mg Q14D (N=6) | Tezepelumab 210 mg Q7D (N=7) | Tezepelumab 700 mg Q28D IV (N=6) | Tezepelumab Total (N=37) | Placebo (N=12)
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Application site dermatitis (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Injection site urticaria (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 2
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 1 | 2 | 3 | 0 | 8 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.